CLINICAL TRIAL: NCT06548178
Title: Neoadjuvant Trastuzumab Deruxtecan (T-DXd) Versus Standard Treatment for Medium-risk HER2-positive Early Breast Cancer: a Randomized, Multi-center Trial (EXTEND)
Brief Title: T-DXd Versus THP for Medium-risk HER2-positive Early Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCHBCC-N077
Record Dates: First submitted 2024-08-04; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): T-DXd (5.4 mg/kg Q3W on Day 1) ×6 cycles.
  Interventions: Drug: T-DXd
- Arm B (Placebo Comparator): Docetaxel (75 mg/m2 Q3W on Day 1) concurrent with trastuzumab (8 mg/kg loading dose followed by 6 mg/kg Q3W on Day 1) and pertuzumab (840 mg loading dose followed by 420 mg Q3W on Day 1) × 6 cycles.
  Interventions: Drug: THP

INTERVENTIONS:
Drug: T-DXd — T-DXd (5.4 mg/kg Q3W on Day 1) ×6 cycles.
  Arms: Arm A
Drug: THP — Docetaxel (75 mg/m2 Q3W on Day 1) concurrent with trastuzumab (8 mg/kg loading dose followed by 6 mg/kg Q3W on Day 1) and pertuzumab (840 mg loading dose followed by 420 mg Q3W on Day 1) × 6 cycles.
  Arms: Arm B

SUMMARY:
This study (EXTEND trial) is a multicentre, interventional, prospective, randomised, open-label, controlled neoadjuvant, phase 2 trial evaluating the efficacy and safety of T-DXd monotherapy vs. standard-of-care docetaxel+ trastuzumab + pertuzumab (THP) in medium-risk (lymph node negative with a primary tumour stage T2) HER2-positive early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥18 years at randomisation
2. Participants with invasive, untreated Locally assessed HER2-positive (IHC 3+ or ISH+) according to ASCO-CAP guidelines (Wolff et al 2018), maximum 6 weeks before registration
3. Clinical stage at presentation (based on mammogram or breast MRI assessment): cT2 (>2cm, ≤5cm ), cN0, M0 as determined by the AJCC staging system, 8th edition (Hortobagyi et al 2017).
4. Written informed consent: Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
5. LVEF ≥ 50% within 28 days before randomisation
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1
7. Adequate organ and bone marrow function within 14 days before randomisation as described: Platelet Count ≥ 100000/mm3; Haemoglobin ≥ 9.0 g/dL; Absolute neutrophil count ≥ 1500/mm3; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN; Total Bilirubin ≤ 1.5×ULN; Serum albumin ≥ 2.5 g/dL; CrCL ≥ 30 mL/min as determined by Cockcroft Gault (using actual body weight). International normalised ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN. All parameters must be the most recent results available.

   Note: Transfusion (red blood cell or platelet) or G-CSF administration is not allowed within 14 days prior to the day on which bone marrow function is assessed, or at any time after this day and prior to C1D1.
8. Adequate treatment washout period before randomisation, defined as: Major Surgery ≥ 4 weeks; Radiation Therapy including palliative stereotactic radiation therapy to chest ≥ 4 weeks; Palliative stereotactic radiation therapy to other anatomic areas including whole brain radiation (see Exclusion Criteria 2) ≥ 2 weeks; Anti-Cancer chemotherapy [Immunotherapy (non-antibody based therapy)], retinoid therapy, hormonal therapy ≥ 3 weeks; Antibody based anti-cancer therapy ≥ 4 weeks; Targeted agents and small molecules ≥ 2 weeks or 5 half-lives, whichever is longer; Nitrosoureas or mitomycin C ≥ 6 weeks; TKIs approved for treatment of NSCLC ≥ 1 week; Chloroquine/Hydroxychloroquine ≥ 14 days; Cell-free and Concentrated Ascites Reinfusion Therapy (CART), peritoneal shunt or drainage of pleural effusion, ascites or pericardial effusion ≥2 weeks prior to screening assessment.
9. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of study treatment.

   Women of childbearing potential are defined as those who are not surgically sterile (i.e., underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
10. Female participants must not donate, or retrieve for their own use, ova from the time of enrolment and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.

Exclusion Criteria:

1. Non-operable breast cancer including inflammatory breast cancer
2. Any previous history of invasive breast cancer
3. Multiple primary malignancies within 3 years, with the exception of

   * adequately resected non-melanoma skin cancer
   * curatively treated in-situ disease
   * other solid tumors curatively treated
4. Any evidence for existing metastatic disease (confirmed by CT Thorax/Abdomen, bone scan, or other methods according to clinical practice
5. Previous or concurrent treatment with cytotoxic agents for any reason (except non-oncological reasons)
6. Concurrent treatment with other experimental drugs and participation in another clinical trial with any investigational drug within 30 days prior to study entry
7. Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study/inadequate organ function
8. Reasons indicating risk of poor compliance
9. Woman of child-bearing potential defined as a woman physiologically capable of becoming pregnant, and not using highly effective methods of contraception during the study treatment and for 3 months after stopping the treatment.
10. Use of oral (oestrogen and progesterone), transdermal, injected, or implanted hormonal methods of contraception as well as hormonal replacement therapy.
11. Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
12. Patients with a medical history of myocardial infarction (MI) within 6 months before randomisation, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrolment to rule out MI.
13. Corrected QT interval (QTcF) prolongation to > 470 msec (females) based on average of the screening triplicate12-lead ECG.
14. History of QT prolongation associated with other medications that required discontinuation of that medication, or any current concomitant medication known to prolong the QT interval and cause TdP.
15. Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.
16. History of (non-infectious) ILD / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
17. Lung criteria:

    * Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
    * Any autoimmune, connective tissue or inflammatory disorders (including Rheumatoid arthritis, Sjogren's and sarcoidosis) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for participants who are included in the study.
    * Prior pneumonectomy (complete)
18. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
19. Active primary immunodeficiency, known uncontrolled active human immunodeficiency virus (HIV) infection or active hepatitis B (hepatitis B virus surface antigen or hepatitis B virus core antibody positive, at screening) or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects should be tested for HIV prior to enrollment if required by local regulations or institutional review board (IRB)/ethics committee (EC).
20. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan or THP standard-of-care treatment.

    Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IMP.
21. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline.

    Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to randomization and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as:
    * Chemotherapy-induced neuropathy
    * Fatigue
    * Residual toxicities from prior IO treatment: Grade 1 or Grade 2 endocrinopathies which may include:

      1. Hypothyroidism/hyperthyroidism
      2. Type 1 diabetes
      3. Hyperglycaemia
      4. Adrenal insufficiency
      5. Adrenalitis
      6. Skin hypopigmentation (vitiligo)
22. Known allergy or hypersensitivity to study treatment (T-DXd) or any of the study drug excipients.
23. History of severe hypersensitivity reactions to other monoclonal antibodies.
24. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.
25. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted upon discussion with the Study Physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 1 year
  pCR rate after neoadjuvant treatment, defined as the proportion of participants who have no evidence by H&E staining of residual invasive disease in the complete resected breast specimen and all sampled regional lymph nodes (ypT0/Tis ypN0) by investigator assessment following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Safety including adverse events (AEs), severe adverse events (SAEs) and adverse events of special interest (AESI). | Up to approximately 1.5 years
  Incidence of AEs, SAE, AESIs (interstitial lung disease, LVEF decrease), AEs resulting in study intervention interruption and discontinuation, etc.
Event-free survival (EFS) rate at 12, 24, 36-month | Up to approximately 3 years
  EFS is defined as time from date of randomisation until disease progression precluding initial surgery, invasive disease recurrence (local, regional, distant, or contralateral), or death from any cause.
Invasive disease-free survival (IDFS) rate at 12, 24, 36-month | Up to approximately 3 years
  IDFS is defined as time from surgery until invasive disease recurrence (local, regional, distant, or contralateral), or death from any cause.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Core 30 Questionnaire (QLQ-C30) score | Up to approximately 3 years
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Individual responses are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome.
EORTC Breast Cancer-Specific QoL Questionnaire (QLQ-BR45) score | Up to approximately 3 years
  The EORTC-QLQ-BR45 is a 45-item questionnaire developed to assess the quality of life of breast cancer patients. Individual responses are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No